CLINICAL TRIAL: NCT01306747
Title: A Randomized Controlled Trial of the Stanford Chronic Pain Self-Management Programme in Danish Chronic Pain Patients
Brief Title: Stanford Chronic Pain Self-Management Programme in Danish Chronic Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: TRYG Foundation (Other); Danish Committee for Health Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACKLE2011
Record Dates: First submitted 2011-02-18; First posted 2011-03-02 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Stanford chronic pain self-management programme; Patient education
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chronic Pain Self-Management (Experimental)
  Interventions: Behavioral: The Stanford Chronic Pain Self-Management Programme
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: The Stanford Chronic Pain Self-Management Programme — The Stanford CPSMP is a patient education program consisting of six 2½ hour weekly sessions. Two trained instructors teach a group of 8-16 persons about managing pain.
  Arms: Chronic Pain Self-Management

SUMMARY:
The effect of the Stanford Chronic Pain Self-Management Programme (CPSMP) is tested in a randomized controlled trial with enrollment of Danish chronic pain patients. A total of 500 chronic pain patients is randomized into either an CPSMP intervention group or a control group.

The CPSMP is brief patient education program consisting of 6 weekly sessions. Two trained instructors teach a group of 8-16 chronic pain patients about managing pain. The instructors are not health professionals but chronic pain patient themselves. The program is highly structured and manualized.

Previous studies have shown beneficial effects of the CPSMP on pain, self-efficacy and well-being. Hence we expect the CPSMP to have an effect on various domains.

1. Symptom reduction - lower self-reported pain in the CPSMP group compared to controls
2. Illness perception - the cpsmp group will differ from controls in illness perception and have higher disease related self-efficacy
3. Sickness behavior - the cpsmp group will have fewer sick days and lower health care utilization (estimated by registerbased data)than controls
4. Quality of life - the cpsmp group will report higher life satisfaction and less social isolation than controls

ELIGIBILITY:
Inclusion Criteria:

* Pain in more than 3 months
* Self-reported pain > 4.99 on 10 point Likert scale
* Age > 18 years old
* Able to understand, speak, and read Danish

Exclusion Criteria:

* Pain related to conditions that the patient are likely to consider more important than pain itself, e.g. pregnancy, cancer in acute phases
* Drug abuse, psychiatric or physical disease that would prevent participation in weekly sessions
* Drug abuse, psychiatric or physical disease that would disturb completion of group sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Decrease in score on the Roland-Morris Disability Questionnaire (Roland & Morris, 1983) | 10 weeks follow-up
Decrease in score on the Roland-Morris Disability Questionnaire (Roland & Morris, 1983) | 6 months follow-up

SECONDARY OUTCOMES:
Increase in score on pain related self-efficacy questionnaire (Lorig et al., 1989) | 10 weeks follow-up
Increase in score on pain related self-efficacy questionnaire (Lorig et al., 1989) | 6 months follow-up
Register-based data on visits to GP after intervention (Danish National Register of Health Care utilization) | 6-months follow-up
Register-based data on use of prescribed drugs after intervention (Danish National Register of Health Care utilization) | 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Per Fink, DMSc, Study Director — Aarhus University Hospital
Locations (1):
- The Research Clinic for Functional Disorders, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Mehlsen M, Hegaard L, Ornbol E, Jensen JS, Fink P, Frostholm L. The effect of a lay-led, group-based self-management program for patients with chronic pain: a randomized controlled trial of the Danish version of the Chronic Pain Self-Management Programme. Pain. 2017 Aug;158(8):1437-1445. doi: 10.1097/j.pain.0000000000000931. PMID 28644822
- See also: Description of the program - In Danish — http://www.patientuddannelse.info/LaerAtTackleKroniskeSmerter.aspx